CLINICAL TRIAL: NCT00002511
Title: PHASE III STUDY OF POST-OPERATIVE EXTERNAL RADIOTHERAPY IN PATHOLOGICAL STAGE T3 N0 PROSTATIC CARCINOMA
Brief Title: Radiation Therapy Compared With No Further Treatment Following Surgery in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-22911; EORTC-22911; EORTC-GU-22911
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells and may be an effective treatment for prostate cancer.

PURPOSE: Randomized phase III trial to compare radiation therapy with no further treatment in treating patients with stage III prostate cancer following radical prostatectomy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare local recurrence rates, acute and late morbidity, overall survival, disease-free survival, and cancer-related survival of patients with pT3 pN0 adenocarcinoma of the prostate randomized following radical prostatectomy to postoperative conventional pelvic irradiation (60 Gy) vs no further treatment until relapse.
* Better define the selective pathologic indications for radiotherapy in patients with pT3 pN0 disease.

OUTLINE: This is a randomized study.

* Arm I: Patients undergo radiotherapy daily, 5 days a week, for 5 weeks, followed by boost radiotherapy for 1-1.4 weeks.
* Arm II: Patients are observed. Local relapse is treated with conventional pelvic radiotherapy.

Patients are followed every 3 months during the first postoperative year, every 6 months until the fifth year, and annually thereafter.

PROJECTED ACCRUAL: A total of 1000 patients will be accrued for this study within 7.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically documented invasive adenocarcinoma of the prostate staged pT3 pN0 after radical prostatectomy

  * Preoperative staging must have been T0-3 N0 M0 based on physical exam, chest x-ray, bone scan, CT or MRI of entire pelvis and abdomen, and serum PSA
  * At least 1 of the following features must be present:

    * Complete capsule invasion (i.e., perforation)
    * Positive surgical margins (microscopic or gross)
    * Seminal vesicle invasion
* Radiotherapy must begin within 16 weeks following surgery, after recovery of urinary function

PATIENT CHARACTERISTICS:

Age:

* 75 and under

Performance status:

* WHO 0-2

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other malignancies

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* No more than 4 months of preoperative hormonal therapy

Radiotherapy:

* Not specified

Surgery:

* Radical prostatectomy required within 12 weeks with recovery of urinary function

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1005 (Actual)
Dates: Start 1992-12; Primary Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Bolla, MD, Study Chair — CHU de Grenoble - Hopital de la Tronche; Hein van Poppel, MD, PhD, Study Chair — University Hospital, Gasthuisberg
Locations (1):
- U.Z. Gasthuisberg, Leuven, Belgium

REFERENCES:
- [Background] Ganswindt U, Stenzl A, Bamberg M, Belka C. Adjuvant radiotherapy for patients with locally advanced prostate cancer--a new standard? Eur Urol. 2008 Sep;54(3):528-42. doi: 10.1016/j.eururo.2008.06.059. Epub 2008 Jun 23. PMID 18602742
- [Background] Gomella LG. Re: identification of patients with prostate cancer who benefit from immediate postoperative radiotherapy: EORTC 22911. Eur Urol. 2008 Apr;53(4):855-6. doi: 10.1016/j.eururo.2008.01.039. PMID 18441534
- [Background] Graefen M. Words of wisdom. Re: Identification of patients with prostate cancer who benefit from immediate postoperative radiotherapy: EORTC 22911. Eur Urol. 2008 Mar;53(3):664-5. doi: 10.1016/j.eururo.2007.12.018. No abstract available. PMID 18365318
- [Result] Bolla M, Van Poppel H, Van Cangh P, et al.: Does post-operative radiotherapy (P-RXT) after radical prostatectomy (Px) improve progression-free survival (PFS) in pT3N0 prostate cancer (PC)? (EORTC 22911). [Abstract] J Clin Oncol 22 (Suppl 14): A-4504, 383, 2004.
- [Result] Bolla M, Van Poppel H, Van Cangh P, et al.: Post-operative radiotherapy (P-RXT) after radical prostatectomy (Px) improves progression-free survival (PFS) in pT3NO prostate cancer (PC) (EORTC 22911). [Abstract] Int J Radiat Oncol Biol Phys 60 (1 Suppl 1): A-93, S186, 2004. Available online. Last accessed January 27, 2005.
- [Result] Bolla M, van Poppel H, Collette L, van Cangh P, Vekemans K, Da Pozzo L, de Reijke TM, Verbaeys A, Bosset JF, van Velthoven R, Marechal JM, Scalliet P, Haustermans K, Pierart M; European Organization for Research and Treatment of Cancer. Postoperative radiotherapy after radical prostatectomy: a randomised controlled trial (EORTC trial 22911). Lancet. 2005 Aug 13-19;366(9485):572-8. doi: 10.1016/S0140-6736(05)67101-2. PMID 16099293
- [Result] Davis JB, Reiner B, Dusserre A, Giraud JY, Bolla M; EORTC. Quality assurance of the EORTC trial 22911. A phase III study of post-operative external radiotherapy in pathological stage T3N0 prostatic carcinoma: the dummy run. Radiother Oncol. 2002 Jul;64(1):65-73. doi: 10.1016/s0167-8140(02)00143-3. PMID 12208577
- [Result] Bolla M, Van Poppel H, Collette L; au nom des groupes genito-urinaire et radiotherapie de l'EORTC. [Preliminary results for EORTC trial 22911: radical prostatectomy followed by postoperative radiotherapy in prostate cancers with a high risk of progression]. Cancer Radiother. 2007 Nov;11(6-7):363-9. doi: 10.1016/j.canrad.2007.09.001. Epub 2007 Oct 10. French. PMID 17931949
- [Result] Van der Kwast TH, Bolla M, Van Poppel H, Van Cangh P, Vekemans K, Da Pozzo L, Bosset JF, Kurth KH, Schroder FH, Collette L; EORTC 22911. Identification of patients with prostate cancer who benefit from immediate postoperative radiotherapy: EORTC 22911. J Clin Oncol. 2007 Sep 20;25(27):4178-86. doi: 10.1200/JCO.2006.10.4067. PMID 17878474
- [Result] Tombal B, Scaillet P, Opsomer R, et al.: Immediate external beam radiation therapy (EBRT) after radical prostatectomy (PCa): long-term influence on QOL, urinary and rectal symptoms. [Abstract] American Urological Association: Annual Meeting, May 20-25, 2006, Atlanta, GA A-1599, 2006.
- [Result] van der Kwast TH, Bolla M, van Poppel H, et al.: Gleason Score and margin status are the strongest predictors for benefit of radiotherapy after radical prostatectomy. [Abstract] American Urological Association: Annual Meeting, May 20-25, 2006, Atlanta, GA A-1391, 2006.
- [Result] van der Kwast TH, Collette L, Van Poppel H, Van Cangh P, Vekemans K, DaPozzo L, Bosset JF, Kurth KH, Schroder FH, Bolla M; European Organisation for Research and Treatment of Cancer Radiotherapy and Genito-Urinary Cancer Groups. Impact of pathology review of stage and margin status of radical prostatectomy specimens (EORTC trial 22911). Virchows Arch. 2006 Oct;449(4):428-34. doi: 10.1007/s00428-006-0254-x. Epub 2006 Aug 29. PMID 16941153
- [Result] Collette L, van Poppel H, Bolla M, van Cangh P, Vekemans K, Da Pozzo L, de Reijke TM, Verbaeys A, Bosset JF, Pierart M; European Organisation for Research and Treatment of Cancer (EORTC) Radiotherapy and Genito-urinary Groups. Patients at high risk of progression after radical prostatectomy: do they all benefit from immediate post-operative irradiation? (EORTC trial 22911). Eur J Cancer. 2005 Nov;41(17):2662-72. doi: 10.1016/j.ejca.2005.06.024. Epub 2005 Oct 11. PMID 16223581
- [Derived] Ritter MA. Commentary on "Postoperative radiotherapy after radical prostatectomy for high-risk prostate cancer: long-term results of a randomised controlled trial (EORTC trial 22911)." Bolla M, van Poppel H, Tombal B, Vekemans K, Da Pozzo L, de Reijke TM, Verbaeys A, Bosset JF, van Velthoven R, Colombel M, van de Beek C, Verhagen P, van den Bergh A, Sternberg C, Gasser T, van Tienhoven G, Scalliet P, Haustermans K, Collette L; European Organisation for Research and Treatment of Cancer, Radiation Oncology and Genito-Urinary Groups. Department of Radiation Oncology, Centre Hospitalier Universitaire A Michallon, Grenoble, France.: Lancet 2012;380(9858):2018-27. doi: 10.1016/S0140-6736(12)61253-7. [Epub 2012 Oct 19]. Urol Oncol. 2014 Apr;32(3):372-3. doi: 10.1016/j.urolonc.2013.09.023. PMID 24679462
- [Derived] Bolla M, van Poppel H, Tombal B, Vekemans K, Da Pozzo L, de Reijke TM, Verbaeys A, Bosset JF, van Velthoven R, Colombel M, van de Beek C, Verhagen P, van den Bergh A, Sternberg C, Gasser T, van Tienhoven G, Scalliet P, Haustermans K, Collette L; European Organisation for Research and Treatment of Cancer, Radiation Oncology and Genito-Urinary Groups. Postoperative radiotherapy after radical prostatectomy for high-risk prostate cancer: long-term results of a randomised controlled trial (EORTC trial 22911). Lancet. 2012 Dec 8;380(9858):2018-27. doi: 10.1016/S0140-6736(12)61253-7. Epub 2012 Oct 19. PMID 23084481